CLINICAL TRIAL: NCT02236039
Title: The Effects of Traffic-Related Air Pollution on Smokers at Risk for Developing COPD
Brief Title: COPD Originates in Polluted Air
Acronym: COPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Christopher Carlsten, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: H14-00821
Record Dates: First submitted 2014-08-11; First posted 2014-09-10 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: COPD
Keywords: Diesel exhaust; Air pollution; Airway responsivness
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Bronchoscopy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Filtered air (Active Comparator): Exposure for 2 hours to filtered air followed by a bronchoscopy 24 hours post exposure.
  Interventions: Procedure: Bronchoscopy
- Diesel exhaust (Experimental): Exposure for 2 hours to diesel exhaust followed by a bronchoscopy 24 hours post exposure.
  Interventions: Procedure: Bronchoscopy

INTERVENTIONS:
Procedure: Bronchoscopy — Bronchoscopy with biopsy sampling, brushings and bronchoalveolar lavage (BAL) 24 hours post exposure.

SUMMARY:
The investigators are investigating the effects of traffic-related diesel exhaust on lung function and the immune system in those at risk for COPD. The individual will be exposed to either filtered air (FA) or carefully controlled levels of diesel exhaust (DE) in our exposure chamber. Post exposure the individual will complete a steady state exercise test. 24h later, a procedure called bronchoscopy (whereby a thin, flexible tube is placed down the throat and into the lungs) will be used so that samples can be collected from the lungs. After 1 month the entire procedure will be repeated with the alternative exposure.

DETAILED DESCRIPTION:
1. Purpose:

   To study the effects of traffic related diesel exhaust on people at risk for developing COPD.
2. Hypotheses:

   Hypothesis 1: An increase in proteins, in the exposed lung and blood, that are associated with the pathophysiology of COPD.

   Hypothesis 2: Air trapping, dyspnea, and impaired exercise tolerance. Such increases will be more pronounced in those with COPD than in control subjects.
3. Justification:

   The use of diesel engines is increasing because they are more fuel-efficient than gasoline engines. However, diesel engines produce different emissions than gasoline engines. Diesel exhaust is emitted from the tailpipe of both "on-road" diesel engine vehicles (diesel cars, buses and trucks) and "non-road" diesel engines (locomotives, marine vessels and some construction equipment). Diesel exhaust consists of both gaseous and particulate air pollutants. People with COPD may be sensitive to air pollution; we would like to know how diesel exhaust (DE) can affects the respiratory and immune systems. We are not expecting that responses will be noticeable to the participant; we are expecting that any responses that may occur will only be detectable through careful examination of cells and tissues (e.g., bronchoalveolar lavage (fluid from lungs), blood). Understanding these subtle changes will help us prevent health problems associated with air pollution in the future.
4. Objectives To provide biological plausibility and deepen mechanistic understanding of the emerging epidemiology suggesting a strong role for air pollution in COPD.
5. Research Methods:

This is a blinded crossover experiment between two conditions (300 µg/m³ diesel exhaust or filtered air), randomized and counter-balanced to order. Data collection for each condition will be separated by a 4-week washout period.

Prior to the exposure participants will: 1) complete some questionnaires, 2) undergo a set of lung function tests (breathing tests), 3) undergo an incremental exercise test and 4) receive a physical exam by the primary investigator. A small sample of blood and spirometry measurements will also be collected for analysis.

After the exposure another series of exercise and lung function tests will be performed. Blood, spirometry measurements, bronchoalveolar lavage (BAL), endobronchial brushings and biopsies will also be collected for examination of cellular, functional and immunological changes influencing the airways.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 40-75 years of age
2. Free of cardiovascular disease
3. Free of insulin-dependent diabetes
4. Study participants must agree to adhere to the following medication intake protocol 24 hours prior to study visits:

   * participants will be asked to withhold:
   * short-acting beta2-agonists (SABAs) for 4 hours prior to testing
   * long-acting beta2-agonists (LABAs) for 12 hours prior to testing if taken in an individual inhaler (different inhaler from inhaled corticosteroid inhaler)
   * LABAs and ICS for 24hrs, if those two medication groups are combined in one inhaler
   * ICS (if taken alone as a mono-therapy, or if taken with either a LABA or SABA, but in two separate inhaler), for 24 hrs.

Overall, we are looking for 15 healthy controls without a history of smoking; 20 individuals with a history of smoking, but who have been non-smokers for at least 6 months prior to study participation; and 15 mild-moderate COPD patients (GOLD I and GOLD II).

Exclusion Criteria:

* Not between the ages of 40-65 years.
* Are pregnant, breast-feeding, or planning to get pregnant in the following 12 months.
* Are currently using inhaled corticosteroids.
* Are allergic to salbutamol, lidocaine, fentanyl or midazolam.
* Are currently participating in another study that involves taking medications.
* Have unstable COPD symptoms.
* Have clinically significant comorbidities (i.e., coronary artery disease).
* Have a history/clinical evidence of asthma.
* Have contraindications to exercise testing.
* Have a body mass index <18.5.
* Regularly use of antihistamines, non-steroidal anti-inflammatories, anticoagulants, acetylsalicylic acid (ASA) or decongestants.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-10-27 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Cytokine pattern | 24 hours
  BAL, BW, and blood cytokines will be assessed at 24h using immunoassays

SECONDARY OUTCOMES:
Gene expression | 24 hours
  BAL, BW, endobronchial brushings and blood will be used for gene expression. RNA will be isolated using RNeasy and supplemented by assessment of promising candidate genes by real-time RT-PCR
Cardiopulmonary function | 1.5 hours
  Cardio pulmonary function will be measured at 1.5 hours post exposure using a cardiopulmonary testing system (Vmax)
Cell culture | 24 hours
  Airway epithelial cells from the endobronchial brushings will be used for non-immortalized cell culture

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Carlsten, MD, MPH, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Behndig AF, Mudway IS, Brown JL, Stenfors N, Helleday R, Duggan ST, Wilson SJ, Boman C, Cassee FR, Frew AJ, Kelly FJ, Sandstrom T, Blomberg A. Airway antioxidant and inflammatory responses to diesel exhaust exposure in healthy humans. Eur Respir J. 2006 Feb;27(2):359-65. doi: 10.1183/09031936.06.00136904. PMID 16452593
- [Background] Hsia CC, Hyde DM, Ochs M, Weibel ER; ATS/ERS Joint Task Force on Quantitative Assessment of Lung Structure. An official research policy statement of the American Thoracic Society/European Respiratory Society: standards for quantitative assessment of lung structure. Am J Respir Crit Care Med. 2010 Feb 15;181(4):394-418. doi: 10.1164/rccm.200809-1522ST. No abstract available. PMID 20130146
- [Background] Gan, W. Q., J. M. FitzGerald, et al. (2013).
- [Background] Mannino DM, Buist AS. Global burden of COPD: risk factors, prevalence, and future trends. Lancet. 2007 Sep 1;370(9589):765-73. doi: 10.1016/S0140-6736(07)61380-4. PMID 17765526
- [Background] Rudell B, Ledin MC, Hammarstrom U, Stjernberg N, Lundback B, Sandstrom T. Effects on symptoms and lung function in humans experimentally exposed to diesel exhaust. Occup Environ Med. 1996 Oct;53(10):658-62. doi: 10.1136/oem.53.10.658. PMID 8943829
- [Background] Schikowski, T., M. Adam, et al. (2014).
- [Background] McCreanor, J., P. Cullinan, et al. (2007).
- [Derived] Ryu MH, Hur SA, Afshar T, Kolmert J, Zurita J, Wheelock CE, Carlsten C. Impact of Short-Term Diesel Exhaust Exposure on Prothrombotic Markers in Chronic Obstructive Pulmonary Disease: A Randomized, Double-Blind, Crossover Study. Ann Am Thorac Soc. 2024 Dec;21(12):1715-1722. doi: 10.1513/AnnalsATS.202311-955OC. PMID 39167788
- [Derived] Yoon M, Ryu MH, Huff RD, Belvisi MG, Smith J, Carlsten C. Effect of traffic-related air pollution on cough in adults with polymorphisms in several cough-related genes. Respir Res. 2022 May 4;23(1):113. doi: 10.1186/s12931-022-02031-8. PMID 35509099
- [Derived] Ryu MH, Afshar T, Li H, Wooding DJ, Orach J, Zhou JS, Murphy S, Lau KSK, Schwartz C, Yuen ACY, Rider CF, Carlsten C. Impact of Exposure to Diesel Exhaust on Inflammation Markers and Proteases in Former Smokers with Chronic Obstructive Pulmonary Disease: A Randomized, Double-blinded, Crossover Study. Am J Respir Crit Care Med. 2022 May 1;205(9):1046-1052. doi: 10.1164/rccm.202104-1079OC. PMID 35202552
- [Derived] Syed N, Ryu MH, Dhillon S, Schaeffer MR, Ramsook AH, Leung JM, Ryerson CJ, Carlsten C, Guenette JA; Canadian Respiratory Research Network. Effects of Traffic-Related Air Pollution on Exercise Endurance, Dyspnea, and Cardiorespiratory Responses in Health and COPD: A Randomized, Placebo-Controlled, Crossover Trial. Chest. 2022 Mar;161(3):662-675. doi: 10.1016/j.chest.2021.10.020. Epub 2021 Oct 23. PMID 34699772
- [Derived] Wooding DJ, Ryu MH, Li H, Alexis NE, Pena O, Carlsten C; Canadian Respiratory Research Network. Acute air pollution exposure alters neutrophils in never-smokers and at-risk humans. Eur Respir J. 2020 Apr 3;55(4):1901495. doi: 10.1183/13993003.01495-2019. Print 2020 Apr. PMID 31806722